CLINICAL TRIAL: NCT02897284
Title: Evaluation of Mindfulness-based Self-care Programs for the Prevention of Burnout Among Primary Care Providers: Psychological, Inflammatory and Epigenetic Effects
Brief Title: Mindfulness for Burnout Prevention in Primary Care Providers
Acronym: Mind-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marcelo Marcos Piva Demarzo, Professor at Preventive Medicine Dept. - Unifesp, Centro Mente Aberta de Mindfulness
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMAMindfulness
Record Dates: First submitted 2016-08-10; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Burnout, Professional
Keywords: Mindfulness-based; Self-care; Health workers; Epigenetics
MeSH Terms: conditions — Burnout, Professional | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness 8 weeks (Experimental): Mindfulness-based intervention with 8 weekly sessions
  Interventions: Behavioral: Mindfulness 8 weeks
- Mindfulness 2 weeks (Active Comparator): Mindfulness-based intervention with 2 weekly sessions
  Interventions: Behavioral: Mindfulness 2 weeks
- Control (No Intervention): waiting list

INTERVENTIONS:
Behavioral: Mindfulness 8 weeks — 8 sessions of mindfulness
  Arms: Mindfulness 8 weeks
Behavioral: Mindfulness 2 weeks — 2 sessions of mindfulness
  Arms: Mindfulness 2 weeks

SUMMARY:
Burnout Syndrome is one of the major challenges for health systems worldwide. This study strives to evaluate the feasibility and effectiveness of an 8- versus 2-week mindfulness-based self-care program on burnout symptoms and psychological and biological variables.

DETAILED DESCRIPTION:
The development of stepped-care interventions allows for the development of new strategies within mindfulness-based approaches, classically described as a weekly two-hour commitment which lasts eight weeks. Such approaches might reach larger and stratified groups, more suitable for usage in Brazilian health-system context. For such evaluations, the investigators will use a 3-arms randomized clinical trial design, with Sociodemographic and Labor variables, such as age, sex, number of offspring, adherence to the program, adherence to the mindfulness practices, Burnout Clinical Subtype Questionnaire -(BCSQ-36), Maslach Burnout Inventory (MBI-GS), Mindfulness Attention Awareness Scale (MAAS), Freiburg Mindfulness Inventory adapted for Brazil (FMI-Br-13), Five-Facet Mindfulness Questionnaire (FFMQ-Br). DNA methylation will be measured by Methylase-reaction, and BDNF (brain-derived neurotrophic factor) will be quantified by ELISA-sandwich. The primary outcome will be the effectiveness of such programs on different clinical subtypes of Burnout symptoms (frenetic, under challenged and worn-out). The secondary outcome will be mindfulness levels, and adherence to the program and to the mindfulness practice, and on inflammation and epigenetic variables.

ELIGIBILITY:
Inclusion Criteria:

* Active Primary Care Providers

Exclusion Criteria:

* Acute disease (physical or mental)
* Schizophrenia or other psychotic symptoms
* Concomitant use of medication causing attentional, cognitive or concentration impairments
* Having practiced mindfulness or other contemplative techniques in the previous 12 months of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
A mindfulness intervention decreases Burnout | up to 2 months of follow-up
  Evaluation of Burnout symptoms through the MBI-GS scale
A mindfulness intervention increases Happiness | up to 2 months of follow-up
  Evaluation of Happiness levels through the PHI (Pemberton) scale

SECONDARY OUTCOMES:
A mindfulness intervention increases Mindfulness | up to 2 months of follow-up
  Evaluation of Mindfulness levels through the MAAS scale
A mindfulness intervention improves Epigenetic | up to 2 months of follow-up
  Evaluation of epigenetic-related activity through Homocysteine levels (Pfeiffer, 1999)
A mindfulness intervention improves Epigenetic (II) | up to 2 months of follow-up
  Evaluation of epigenetic-related activity through Cysteine levels (Pfeiffer, 1999)
A mindfulness intervention improves Epigenetic (III) | up to 2 months of follow-up
  Evaluation of epigenetic-related activity through Methylase Reaction (Radiomarking of methyl groups)
A mindfulness intervention improves Inflammation | up to 2 months of follow-up
  Evaluation of inflammation-related activity through seric Brain-Derived Neurotrophic Factor - BDNF- (ELISA-Sandwich)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MP Demarzo, MD, PhD, Principal Investigator — Mente Aberta - Brazilian Center for Mindfulness and Health Promotion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barros VV. Evidências de validade da Escala de Atenção e Consciência Plenas (MAAS) e do Questionário das Facetas de Mindfulness (FFMQ-BR) entre usuários de tabaco e população geral [dissertação]. Juiz de Fora (MG): Universidade Federal de Juiz de Fora; 2013.
- [Background] Bower P, Gilbody S. Stepped care in psychological therapies: access, effectiveness and efficiency. Narrative literature review. Br J Psychiatry. 2005 Jan;186:11-7. doi: 10.1192/bjp.186.1.11. PMID 15630118
- [Background] Garcia Campayo J. [The practice of "being attentive" (mindfulness) in medicine. Impact on patients and professionals]. Aten Primaria. 2008 Jul;40(7):363-6. doi: 10.1157/13124130. No abstract available. Spanish. PMID 18620639
- [Background] Cavanagh K, Strauss C, Cicconi F, Griffiths N, Wyper A, Jones F. A randomised controlled trial of a brief online mindfulness-based intervention. Behav Res Ther. 2013 Sep;51(9):573-8. doi: 10.1016/j.brat.2013.06.003. Epub 2013 Jun 28. PMID 23872699
- [Background] Coyle D, Doherty G. Stepped care and mental health technologies, en ECCE 2010 workshop on Cognitive Engineering for Technology in Mental Health Care and Rehabilitation, pp. 99-102, 2010.
- [Background] Demarzo MMP. Meditação aplicada à saúde. Programa Atualização em Med Família e Comunidade. 6th ed. Porto ALegre-RS: Artmed; 2011;6(1):1-18.
- [Background] Demarzo MM, Andreoni S, Sanches N, Perez S, Fortes S, Garcia-Campayo J. Mindfulness-based stress reduction (MBSR) in perceived stress and quality of life: an open, uncontrolled study in a Brazilian healthy sample. Explore (NY). 2014 Mar-Apr;10(2):118-20. doi: 10.1016/j.explore.2013.12.005. Epub 2013 Dec 18. No abstract available. PMID 24607079
- [Background] Epstein RM, Krasner MS. Physician resilience: what it means, why it matters, and how to promote it. Acad Med. 2013 Mar;88(3):301-3. doi: 10.1097/ACM.0b013e318280cff0. PMID 23442430
- [Background] Gluck TM, Maercker A. A randomized controlled pilot study of a brief web-based mindfulness training. BMC Psychiatry. 2011 Nov 8;11:175. doi: 10.1186/1471-244X-11-175. PMID 22067058
- [Background] Hesser H, Gustafsson T, Lunden C, Henrikson O, Fattahi K, Johnsson E, Zetterqvist Westin V, Carlbring P, Maki-Torkko E, Kaldo V, Andersson G. A randomized controlled trial of Internet-delivered cognitive behavior therapy and acceptance and commitment therapy in the treatment of tinnitus. J Consult Clin Psychol. 2012 Aug;80(4):649-61. doi: 10.1037/a0027021. Epub 2012 Jan 16. PMID 22250855
- [Background] Hirayama MS. Freiburg Mindfulness Inventory: Adaptação cultural e validação para a língua portuguesa no Brasil. [tese]. Campinas (SP): Universidade estadual de Campinas, 2014.
- [Background] Hirayama MS, Milani D, Rodrigues RC, Barros NF, Alexandre NM. [The perception of behavior related to mindfulness and the Brazilian version of the Freiburg Mindfulness Inventory]. Cien Saude Colet. 2014 Sep;19(9):3899-914. doi: 10.1590/1413-81232014199.12272013. Portuguese. PMID 25184595
- [Background] Irving JA, Dobkin PL, Park J. Cultivating mindfulness in health care professionals: a review of empirical studies of mindfulness-based stress reduction (MBSR). Complement Ther Clin Pract. 2009 May;15(2):61-6. doi: 10.1016/j.ctcp.2009.01.002. Epub 2009 Feb 28. PMID 19341981
- [Background] Franco Justo C. [Reducing stress levels and anxiety in primary-care physicians through training and practice of a mindfulness meditation technique]. Aten Primaria. 2010 Nov;42(11):564-70. doi: 10.1016/j.aprim.2009.10.020. Epub 2010 Feb 2. Spanish. PMID 20129713
- [Background] Keng SL, Smoski MJ, Robins CJ. Effects of mindfulness on psychological health: a review of empirical studies. Clin Psychol Rev. 2011 Aug;31(6):1041-56. doi: 10.1016/j.cpr.2011.04.006. Epub 2011 May 13. PMID 21802619
- [Background] Kerrigan D, Johnson K, Stewart M, Magyari T, Hutton N, Ellen JM, Sibinga EM. Perceptions, experiences, and shifts in perspective occurring among urban youth participating in a mindfulness-based stress reduction program. Complement Ther Clin Pract. 2011 May;17(2):96-101. doi: 10.1016/j.ctcp.2010.08.003. Epub 2010 Sep 16. PMID 21457899
- [Background] Krusche A, Cyhlarova E, King S, Williams JM. Mindfulness online: a preliminary evaluation of the feasibility of a web-based mindfulness course and the impact on stress. BMJ Open. 2012 May 21;2(3):e000803. doi: 10.1136/bmjopen-2011-000803. Print 2012. PMID 22614170
- [Background] Ljotsson B, Falk L, Vesterlund AW, Hedman E, Lindfors P, Ruck C, Hursti T, Andreewitch S, Jansson L, Lindefors N, Andersson G. Internet-delivered exposure and mindfulness based therapy for irritable bowel syndrome--a randomized controlled trial. Behav Res Ther. 2010 Jun;48(6):531-9. doi: 10.1016/j.brat.2010.03.003. Epub 2010 Mar 16. PMID 20362976
- [Background] Martin Asuero A, Rodriguez Blanco T, Pujol-Ribera E, Berenguera A, Moix Queralto J. [Effectiveness of a mindfulness program in primary care professionals]. Gac Sanit. 2013 Nov-Dec;27(6):521-8. doi: 10.1016/j.gaceta.2013.04.007. Epub 2013 May 28. Spanish. PMID 23721869
- [Background] Mateen FJ, Dorji C. Health-care worker burnout and the mental health imperative. Lancet. 2009 Aug 22;374(9690):595-7. doi: 10.1016/S0140-6736(09)61483-5. No abstract available. PMID 19699996
- [Background] Monshat K, Castle DJ. Mindfulness training: an adjunctive role in the management of chronic illness? Med J Aust. 2012 May 21;196(9):569-71. doi: 10.5694/mja11.10974. PMID 22621147
- [Background] McCabe Ruff K, Mackenzie ER. The role of mindfulness in healthcare reform: a policy paper. Explore (NY). 2009 Nov-Dec;5(6):313-23. doi: 10.1016/j.explore.2009.10.002. No abstract available. PMID 19913756
- [Background] Montero-Marin J, Araya R, Blazquez BO, Skapinakis P, Vizcaino VM, Garcia-Campayo J. Understanding burnout according to individual differences: ongoing explanatory power evaluation of two models for measuring burnout types. BMC Public Health. 2012 Oct 30;12:922. doi: 10.1186/1471-2458-12-922. PMID 23110723
- [Background] Montero-Marin J, Garcia-Campayo J. A newer and broader definition of burnout: validation of the "Burnout Clinical Subtype Questionnaire (BCSQ-36)". BMC Public Health. 2010 Jun 2;10:302. doi: 10.1186/1471-2458-10-302. PMID 20525178
- [Background] Moreira Dde S, Magnago RF, Sakae TM, Magajewski FR. [Prevalence of burnout syndrome in nursing staff in a large hospital in south of Brazil]. Cad Saude Publica. 2009 Jul;25(7):1559-68. doi: 10.1590/s0102-311x2009000700014. Portuguese. PMID 19578577
- [Background] Morse G, Salyers MP, Rollins AL, Monroe-DeVita M, Pfahler C. Burnout in mental health services: a review of the problem and its remediation. Adm Policy Ment Health. 2012 Sep;39(5):341-52. doi: 10.1007/s10488-011-0352-1. PMID 21533847
- [Background] Morris ME, Kathawala Q, Leen TK, Gorenstein EE, Guilak F, Labhard M, Deleeuw W. Mobile therapy: case study evaluations of a cell phone application for emotional self-awareness. J Med Internet Res. 2010 Apr 30;12(2):e10. doi: 10.2196/jmir.1371. PMID 20439251
- [Background] Nakamura E. O Método Etnográfico em Pesquisas na Área da Saúde: uma reflexão antropológica Saúde Soc. São Paulo, v.20, n.1, p.95-103, 2011
- [Background] Nakao M. Epigenetics: interaction of DNA methylation and chromatin. Gene. 2001 Oct 31;278(1-2):25-31. doi: 10.1016/s0378-1119(01)00721-1. PMID 11707319
- [Background] Nunes DFS, de Souza WL, do Prado AF, Demarzo MMP. Designing an ubiquitous computing environment for monitoring physical activity. 2012 25th IEEE International Symposium on Computer-Based Medical Systems (CBMS) [Internet]. IEEE; 2012 [cited 2013 Aug 10]. p. 1-6. Available from: http://ieeexplore.ieee.org/lpdocs/epic03/wrapper.htm?arnumber=6266383
- [Background] Pfeiffer CM, Huff DL, Gunter EW. Rapid and accurate HPLC assay for plasma total homocysteine and cysteine in a clinical laboratory setting. Clin Chem. 1999 Feb;45(2):290-2. No abstract available. PMID 9931056
- [Background] Queiroz DT, Vall J, Souza AMA, Vieira NFC. Observação participante na pesquisa qualitativa: conceitos e aplicações na área da saúde. R Enferm UERJ,15(2):276-83, 2007.
- [Background] Richards DA. Stepped care: a method to deliver increased access to psychological therapies. Can J Psychiatry. 2012 Apr;57(4):210-5. doi: 10.1177/070674371205700403. PMID 22480585
- [Background] Rodriguez-Dorantes M, Tellez-Ascencio N, Cerbon MA, Lopez M, Cervantes A. [DNA methylation: an epigenetic process of medical importance]. Rev Invest Clin. 2004 Jan-Feb;56(1):56-71. Spanish. PMID 15144044
- [Background] Silva ATC da, Menezes PR. Esgotamento profissional e transtornos mentais comuns em agentes comunitários de saúde. Rev Saude Publica [Internet]. Faculdade de Saúde Pública da Universidade de São Paulo; 2008 Oct [cited 2013 Aug 9];42(5):921-9. Available from: http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0034-89102008000500019&lng=en&nrm=iso&tlng=pt
- [Background] Trigo TR, Teng CT, Hallak JEC. Síndrome de burnout ou estafa profissional e os transtornos psiquiátricos. Rev Psiquiatr Clínica [Internet]. Faculdade de Medicina da Universidade de São Paulo; 2007 [cited 2013 Aug 9];34(5):223-33. Available from: http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0101-60832007000500004&lng=pt&nrm=iso&tlng=pt
- [Background] Tucunduva LT, Garcia AP, Prudente FV, Centofanti G, de Souza CM, Monteiro TA, Vince FA, Samano ES, Goncalves MS, Del Giglio A. [Incidence of the burnout syndrome among Brazilian cancer physicians]. Rev Assoc Med Bras (1992). 2006 Mar-Apr;52(2):108-12. doi: 10.1590/s0104-42302006000200021. Epub 2006 Jun 1. Portuguese. PMID 16767336
- [Background] Zernicke KA, Campbell TS, Speca M, McCabe-Ruff K, Flowers S, Dirkse DA, Carlson LE. The eCALM Trial-eTherapy for cancer appLying mindfulness: online mindfulness-based cancer recovery program for underserved individuals living with cancer in Alberta: protocol development for a randomized wait-list controlled clinical trial. BMC Complement Altern Med. 2013 Feb 16;13:34. doi: 10.1186/1472-6882-13-34. PMID 23414206
- [Background] Wolffe AP, Matzke MA. Epigenetics: regulation through repression. Science. 1999 Oct 15;286(5439):481-6. doi: 10.1126/science.286.5439.481. PMID 10521337